CLINICAL TRIAL: NCT04891601
Title: Randomised Controlled Trial, Compare Mesh and Combined Mesh and Darn Repair in the Treatment of Adults Inguinal Hernia
Brief Title: Mesh Alone VS Combined Mesh and Darn in the Management of Primary Inguinal Hernia in Adult Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jabir Ibn Hayyan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hernia
Record Dates: First submitted 2021-03-08; First posted 2021-05-18 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-05

CONDITIONS: Inguinal Hernia
Keywords: Adult inguinal hernia; Mesh; Darn repair; Hernia repair techinques; Primary inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group II MA Mesh alone repair (Active Comparator): patient use mesh alone as treatment of inguinal hernia
  Interventions: Procedure: polypropelene mesh
- Group I CMD Combined Mesh & darn (Active Comparator): patients utilize both mesh and darn repair
  Interventions: Procedure: polypropelene mesh

INTERVENTIONS:
Procedure: polypropelene mesh — compare use mesh alone or combined mesh and darn repair

SUMMARY:
A prospective randomized study involved 228 individuals with primary inguinal hernia, operated in our departments, between January 2015 to February 2018. The duration of hospital stay, operative time, duration of returning to routine activities, postsurgical sequels and recurrence rates estimated. We randomly allocated it into two groups: mesh repair was applied to 166 patients (Group 1) and combined both mesh, and darn repair applied to 162 patients (Group 2).

DETAILED DESCRIPTION:
Background In spite of the era of laparoscopy still, open repair in primary inguinal hernia is currently the most commonly performed general surgical operation. To evaluate whether the combined darn repair plus Lichtenstein compare Lichtenstein repair alone in the treatment of inguinal hernias regarding postoperative complication and recurrence.

Materials and methods:

A prospective randomized study involved with 218 patients with primary inguinal hernia, operated in our departments, between 2015 and 2018. The duration of the operation time, hospitalization, and time to return to daily activities and postoperative complication and recurrence rates were evaluated. We randomly allocated into two groups: Lichtenstein repair was applied to 169 patients (Group 1), and combined both modified darn repair plus Lichtenstein repair was applied to 160 patients (Group 2).

Results:

The average follow-up period was 48 months. For the alone Lichtenstein procedure, the average duration of operation was 62 min; the average time to return to routine activities was 21 days. The number of patients with postoperative complications was 12 (11.3 %), and the number of patients with recurrence was 1 (0. 9%). For darn repair plus Lichtenstein procedure, the average duration of operation was 72 min; the time to return to daily activities was 21days. The number of patients with postoperative complication was 13 (11.6%), and no recurrences were noted. The hospitalization time of the groups was similar.

Conclusion:

Two-year follow-up, combined mesh and darn better than mesh alone in recurrence rate, both had the same postoperative complication, hospitalization time and return to routine activity.

ELIGIBILITY:
Inclusion Criteria:

* primary hernia
* male

Exclusion Criteria:

* Female
* bilateral
* recurrent hernia

Ages: 16 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | two to four year
  follow up
Post operative complications | two to four year
  record complication
Post operative pain | two to four year
  Visual Analog Score for pain

IPD SHARING:
Plan to Share IPD: Undecided
Yes